CLINICAL TRIAL: NCT07273552
Title: Efficacy of Root Torque Control in Adult Non-extraction Spacing Cases Treated With Directly 3D Printed Clear Aligners: a Cone Beam Computed Tomography Study
Brief Title: Root Torque Control in Cases Treated With Direct Printed Aligners
Acronym: CBCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Collaborators: British University In Egypt (Other); Beni-Suef University (Other)
Responsible Party: Principal Investigator, rim fathalla, Rim Mohamed Fathalla Eissa, Suez Canal University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #REC-FDBSU/08052025-01/AR
Record Dates: First submitted 2025-11-19; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Effect of Direct Printed Aligners on Root Torque
Keywords: Direct printed aligners torque

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with spacing (Experimental): Patients will receive direct printed aligners to treat the spacing
  Interventions: Other: Direct printed aligners

INTERVENTIONS:
Other: Direct printed aligners — After intraoral scanning and CBCT taking, patients will receive Direct printed aligners, each set will be changed after 10 days, till the patients finish their treatment, then a post-CBCT scan will be taken from each patient.

SUMMARY:
This study aims to three-dimensionally evaluate the efficiency of direct 3D printed aligners in achieving the planned root torque by using CBCT and to assess the associated bone thickness changes and root resorption.

DETAILED DESCRIPTION:
Participants will be recruited from the Faculty of Dentistry, Beni Suef, Suez Canal, and British Universities. All subjects will be informed of the treatment procedures and will sign a consent form.

the minimum total required sample size (n) was found to be (14) cases. The sample size was calculated using R statistical analysis software version 4.5.0 for Windows[11].

Methodology:

* Cone beam computed tomography scans will be done before treatment (T0).
* Intraoral scanning of the patients will be performed by using an intraoral scanner to obtain pre-treatment digital models of the upper and lower arches. The treatment plan will be set up, and the aligners will be 3D printed.
* The patient will be instructed to immerse the aligners in warm water before inserting them into the mouth to soften them and improve their fit. The patient will be instructed to change the aligners every week.
* At the end of orthodontic treatment (within 9 months - 2 years after the beginning of the treatment), a post-treatment CBCT scan will be obtained (T1)
* The achieved torque movement of the upper and lower incisors will be calculated by evaluated the pre and post CBCT scans taking the difference between T0 and T1.
* The difference between achieved and predicted torque movement (DAPM) will be obtained, and the efficiency will be calculated by dividing the achieved movement / predicted movement X 100 %
* The labial and palatal bone thickness and root length of the upper and lower incisors will be measured at T0 and T1 by using the pre and post cone-beam computed tomography, and the difference will be calculated.

The results will be obtained and statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18- 45 years old.
2. Non- extraction treatment.
3. Angle Class I or Class II dental malocclusion with generalized or localized anterior spacing.
4. Normal probing depth.

Exclusion Criteria:

1. Active periodontal disease.
2. Crowding cases.
3. Systemic diseases or medications that alter bone metabolism or tooth movement.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the efficacy of direct 3D printed aligners in achieving the planned root torque of upper and lower incisors . | 9-12 months

SECONDARY OUTCOMES:
Change in the bone thickness (measured in mm) around the upper and lower incisors associated with the achieved root torque. | 9-12 months
Assessment of amount of root resorption (measured in mm) of upper and lower incisors associated with root torque. | 9-12 months

CONTACTS AND LOCATIONS:
Overall Officials: Rim M Fathalla, PhD of Orthodontics, Principal Investigator — Suez Canal University
Locations (3):
- Egypt (3):
  - Beni-Suef University, Banī Suwayf
  - British University in Egypt, Cairo
  - Suez Canal University, Ismailia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Iglesias-Linares A, Sonnenberg B, Solano B, Yanez-Vico RM, Solano E, Lindauer SJ, Flores-Mir C. Orthodontically induced external apical root resorption in patients treated with fixed appliances vs removable aligners. Angle Orthod. 2017 Jan;87(1):3-10. doi: 10.2319/02016-101.1. Epub 2016 Aug 9. PMID 27504821
- [Result] Li Y, Deng S, Mei L, Li Z, Zhang X, Yang C, Li Y. Prevalence and severity of apical root resorption during orthodontic treatment with clear aligners and fixed appliances: a cone beam computed tomography study. Prog Orthod. 2020 Jan 6;21(1):1. doi: 10.1186/s40510-019-0301-1. PMID 31903505
- [Result] Lacruz RS, de Castro JM, Martinon-Torres M, O'Higgins P, Paine ML, Carbonell E, Arsuaga JL, Bromage TG. Facial morphogenesis of the earliest europeans. PLoS One. 2013 Jun 6;8(6):e65199. doi: 10.1371/journal.pone.0065199. Print 2013. PMID 23762314
- [Result] Zhang XJ, He L, Guo HM, Tian J, Bai YX, Li S. Integrated three-dimensional digital assessment of accuracy of anterior tooth movement using clear aligners. Korean J Orthod. 2015 Nov;45(6):275-81. doi: 10.4041/kjod.2015.45.6.275. Epub 2015 Nov 20. PMID 26629473
- [Result] Sfondrini MF, Gandini P, Castroflorio T, Garino F, Mergati L, D'Anca K, Trovati F, Scribante A. Buccolingual Inclination Control of Upper Central Incisors of Aligners: A Comparison with Conventional and Self-Ligating Brackets. Biomed Res Int. 2018 Nov 29;2018:9341821. doi: 10.1155/2018/9341821. eCollection 2018. PMID 30627583
- [Result] Tartaglia GM, Mapelli A, Maspero C, Santaniello T, Serafin M, Farronato M, Caprioglio A. Direct 3D Printing of Clear Orthodontic Aligners: Current State and Future Possibilities. Materials (Basel). 2021 Apr 5;14(7):1799. doi: 10.3390/ma14071799. PMID 33916462